CLINICAL TRIAL: NCT03196154
Title: Cross-Sectional Study on Association Between the Estimation of Insulin Resistance and Beta Cell Function Through Homeostasis Model Assessment With HbA1C Among Oral Anti-Diabetics Treatment Non-Responders
Brief Title: Association Between Insulin Resistance and Beta Cell Function With HbA1C in Diabetics
Acronym: InsuReB
Status: Completed | Type: Observational
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Aylwin Lim Ming Wee, Research Pharmacist, Clinical Research Centre, Malaysia
Other Study IDs: NMRR-17-122-33927
Record Dates: First submitted 2017-06-19; First posted 2017-06-22 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Homeostasis Model Assessment; Insulin Resistance; Beta Cell Function; Liquid Chromatography Tandem Mass Spectrometry
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metformin: Patients who are on either metformin 2g per day or metformin extended release 2g per day. Subject will be required to fast overnight. Fasting insulin levels and plasma drug levels will be measured.
  Interventions: Diagnostic Test: Fasting insulin level; Diagnostic Test: Plasma drug level
- Metformin + Gliclazide: Patient who are on both metformin 2g per day or metformin extended release 2g per day and gliclazide 320mg per day or gliclazide modified release 120mg per day. Subject will be required to fast overnight. Fasting insulin levels and plasma drug levels will be measured.
  Interventions: Diagnostic Test: Fasting insulin level; Diagnostic Test: Plasma drug level

INTERVENTIONS:
Diagnostic Test: Fasting insulin level — Fasting insulin and C-peptide level measured using LCMS which is then used to calculate the insulin resistance and beta cell function using homeostasis model assessment
Diagnostic Test: Plasma drug level — Plasma trough level of metformin and gliclazide will be measured using LCMS to ensure true compliance.

SUMMARY:
Progression of T2DM is widely accepted to be contributed by two main components: beta cell function deterioration where insulin secretion is impaired and insulin resistance where insulin physiological response is reduced. Insulin resistance and beta cell function will be estimated through a mathematical model, homeostasis model assessment. Fasting insulin and C-peptide will be measured using liquid chromatography tandem mass spectrometry. Insulin resistance and beta cell function is then compared with the glycaemic control, HbA1C.

DETAILED DESCRIPTION:
Primary objective

• To investigate the association between the estimation of insulin resistance and beta cell function through homeostasis model assessment with HbA1C among oral anti-diabetics treatment non-responder.

Secondary Objectives

* To compare the insulin resistance and beta cell function between the OAD treatment responders (negative control) and non-responders
* To investigate the relationship between plasma level of metformin and gliclazide with the estimation of beta cell function and insulin resistance
* To identify the proportion of patients with high insulin resistance and proportion of patients with low beta cell function
* To identify difference in insulin resistance and beta cell function of different ethnic groups in Sarawak
* To compare insulin resistance with cardiovascular disease risk using Framingham Risk Score and ASCVD risk estimation

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed to have T2DM, currently treated with oral anti-diabetics agents (either on maximum dose of Metformin only or with maximum dose of Gliclazide) for at least 3 months with no change in medications and dosage during the period of 3 months

Exclusion Criteria:

* Patient that is on exogenous insulin, is on hormone replacement therapy or any steroids medications, with renal impairment with creatinine clearance less than 30ml/min and unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All T2DM patients under Sarawak General Hospital, Sarawak Heart Centre, Tanah Puteh Health Clinic, Jalan Masjid Health Clinic and Petra Jaya Health Clinic follow up during the period 3 July 2017 until 30 March 2018
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
HOMA estimation of insulin resistance and beta cell function | 1 day
  Insulin resistance and beta cell function is estimated through homeostasis model assessment
HbA1C | 1 day
  Glycaemic control of subjects assessed through HbA1C

SECONDARY OUTCOMES:
Medication adherence | 1 day
  Assessed using Malaysian Medication Adherence Scale
Plasma metformin level | 1 day
  Measured using LCMS
Plasma gliclazide level | 1 day
  Measured using LCMS
Cardiovascular risk estimation | 1 day
  Framingham risk score and ASCVD risk estimation

CONTACTS AND LOCATIONS:
Overall Officials: Aylwin Ming Wee Lim, Principal Investigator — Clinical Research Centre, Malaysia
Locations (1):
- Clinical Research Centre, Sarawak General Hospital, Kuching, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No